CLINICAL TRIAL: NCT05471440
Title: SWITCH ON: Analysing the Immunogenicity of Additional Booster Vaccinations in Healthcare Workers. A Multicenter, Randomised, Controlled Trial
Brief Title: SWITCH ON: Analysing the Immunogenicity of Additional Booster Vaccinations in HCW
Acronym: SWITCHON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Leiden University Medical Center (Other); University Medical Center Groningen (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Hugo van der Kuy, Head Department Clinical Pharmacy/ Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MEC-2022-0462; 2022-002560-73 (EudraCT Number)
Record Dates: First submitted 2022-07-17; First posted 2022-07-22 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Covid-19 Vaccination
Keywords: Covid-19; Boost
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: A multicenter, randomized, controlled trial comparing immune responses 7 and 28 days after an additional COVID-19 booster vaccination between Janssen and mRNA primed HCWs to describe the immune response in a cohort representative of the Dutch population, in order to eventually provide data for Dutch policy makers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Direct boost mRNA (Active Comparator): Participants will be randomised into a direct boost group (DB; i.e end of August) or a post-poned boost group (PPB; i.e 3-4 months later) group after stratification for priming (mRNA versus Janssen). The immune response will be measured at start of the study (visit 1, all participants) and 0, 7, 28 and 84 days after boost.
  Interventions: Drug: Direct boost mRNA
- Direct boost adeno (Active Comparator): Participants will be randomised into a direct boost group (DB; i.e end of August) or a post-poned boost group (PPB; i.e 3-4 months later) group after stratification for priming (mRNA versus Janssen). The immune response will be measured at start of the study (visit 1, all participants) and 0, 7, 28 and 84 days after boost.
  Interventions: Drug: Direct boost adeno
- Post-poned boost mRNA (Active Comparator): Participants will be randomised into a direct boost group (DB; i.e end of August) or a post-poned boost group (PPB; i.e 3-4 months later) group after stratification for priming (mRNA versus Janssen). The immune response will be measured at start of the study (visit 1, all participants) and 0, 7, 28 and 84 days after boost.
  Interventions: Drug: Post-poned boost mRNA
- Post-poned boost adeno (Active Comparator): Participants will be randomised into a direct boost group (DB; i.e end of August) or a post-poned boost group (PPB; i.e 3-4 months later) group after stratification for priming (mRNA versus Janssen). The immune response will be measured at start of the study (visit 1, all participants) and 0, 7, 28 and 84 days after boost.
  Interventions: Drug: Post-poned boost adeno

INTERVENTIONS:
Drug: Direct boost mRNA — Participants will be boosted with a covid-19 vaccin after priming with mRNA
  Arms: Direct boost mRNA
Drug: Direct boost adeno — Participants will be boosted with a covid-19 vaccin after priming with adeno
  Arms: Direct boost adeno
Drug: Post-poned boost mRNA — Participants will be boosted with a covid-19 vaccin after priming with mRNA
  Arms: Post-poned boost mRNA
Drug: Post-poned boost adeno — Participants will be boosted with a covid-19 vaccin after priming with adeno
  Arms: Post-poned boost adeno

SUMMARY:
Eighty percent of the Dutch population has completed a primary COVID-19 vaccination regimen, and 60% of the population received a booster vaccination. Waning immunity, combined with the emergence of antigenically distinct SARS-CoV-2 variants, has led to the consideration of additional booster vaccinations in the Dutch population by autumn 2022. However, despite efforts of the Dutch policymakers, the public's willingness to repeatedly receive COVID-19 booster vaccinations is declining. This is mainly due to a reduced burden of disease by COVID-19, fewer hospitalizations, and fewer deaths. However, population immunity might be one of the major factors responsible for this reduced burden of disease, possibly emphasizing the need for booster vaccinations. In this proposal we will address an important question asked by policymakers: "Are booster vaccinations in autumn recommended for the healthy population?"

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give written informed consent for participation in the trial.
2. Adult (male/female) between 18 and 65 years old
3. Sufficient level of the Dutch language to undertake all study requirements

Exclusion Criteria:

1. Adults younger than 18 or older than 65 years.
2. Adults primed with another vaccine than Janssen, Moderna or Pfizer.
3. History of allergic reactions likely to be exacerbated by any component of study vaccines (e.g. hypersensitivity to the active substance or any of the SmPC-listed ingredients of the Janssen/Pfizer/Moderna vaccine).
4. Adults that are pregnant.
5. Currently being treated for cancer.
6. Severe kidney failure or dialyses dependent.
7. Status after organ-, stem cell- or bone marrow transplantation.
8. Use of immunosuppressant's.
9. Epilepsy.
10. HIV.
11. Bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding of bruising following IM injections of vene puncture.
12. Continuous use of anticoagulants, such as coumarins (e.g. acenocoumarol) or novel oral anticoagulants (i.e. apixaban, dabigatran etc).
13. Participants who are currently participating in another research trial.
14. All regular contra-indications of the vaccines will be applied.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2022-08-20 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Is there an increase in antibody levels between day of boost and 28 days after boosting HCW that were initially primed with either the Janssen or an mRNA-based vaccine? | 28 days
  Outcome: Level and fold change of antibodies determined by a quantitative IgG assay comparing the Janssen primed and mRNA-based primed HCW.
Does booster vaccination lead to a rapid secondary recall response, indicative of immunological memory? | 28 days
  Outcome: Level and fold change of antibodies and T-cell responses determined by a quantitative IgG assay and whole blood IFNγ release assay, respectively, comparing day 7 and 28 post-boost.

SECONDARY OUTCOMES:
What is the difference in booster immunogenicity comparing a direct boost with a postponed boost? | 28 days
  Outcome: Level of antibodies and T-cell responses 7 and 28 days post boost in DB versus PPB group.
What is the breadth of the immune responses after booster vaccination? | 28 days
  Outcome: PRNT against relevant variants in a random selection of study participants.
What is the predictive value of immune responses on day 7 post boost? | 28 days
  Outcome: Correlation between antibodies and T-cell responses on day 7 and 28 post boost in % of the 28 day response for both level of antibodies and T-cell responses
What is the difference in reactogenicity 7 days after boost comparing the Janssen and mRNA primed HCW? | 7 days
  Outcome: Adverse events (AE) first 7 days after an additional boost between Janssen and mRNA primed HCW.
Initial examination of breakthrough infections before and during study period | 1 year
  Outcome: Database of breakthrough infections in included participants based on positive PCR, self-reported positive lateral flow test, or detection of N-specific antibodies.

OTHER OUTCOMES:
Gene expression profiles associated with recall response (PAXgene tube) | 28 days
SARS-CoV-2-specific T-cell responses | 28 days
  PBMC, assessed by activation-induced marker assay and / or TCRbeta sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Hugo van der Kuy, PharmD, Principal Investigator — Erasmus MC, Rotterdam
Locations (4):
- Netherlands (4):
  - AmsterdamUMC, Amsterdam
  - UMCG, Groningen
  - LUMC, Leiden
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared upon a reasonable request to the PI of the study.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: These data will become available 3 months after the start of the trial
Access Criteria: a reasonable request

REFERENCES:
- [Derived] Tan NH, Lafeber M, Sablerolles RSG, Veerman Roders I, van de Hoef A, van Grafhorst K, Visser LG, Postma DF, Goorhuis A, Rietdijk WJR, van der Kuy PHM. Evaluation of a group-based online informed consent conversation (eConsent) in participants from a low-risk vaccination clinical trial. Trials. 2024 Aug 7;25(1):528. doi: 10.1186/s13063-024-08367-4. PMID 39107860
- [Derived] Tan NH, Geers D, Sablerolles RSG, Rietdijk WJR, Goorhuis A, Postma DF, Visser LG, Bogers S, van Dijk LLA, Gommers L, van Leeuwen LPM, Boerma A, Nijhof SH, van Dort KA, Koopmans MPG, Dalm VASH, Lafeber M, Kootstra NA, Huckriede ALW, van Baarle D, Zaeck LM, GeurtsvanKessel CH, de Vries RD, van der Kuy PHM; SWITCH ON Research Group. Immunogenicity of bivalent omicron (BA.1) booster vaccination after different priming regimens in health-care workers in the Netherlands (SWITCH ON): results from the direct boost group of an open-label, multicentre, randomised controlled trial. Lancet Infect Dis. 2023 Aug;23(8):901-913. doi: 10.1016/S1473-3099(23)00140-8. Epub 2023 Apr 21. PMID 37088096
- [Derived] Tan NH, Sablerolles RSG, Rietdijk WJR, Goorhuis A, Postma DF, Visser LG, Bogers S, Geers D, Zaeck LM, Koopmans MPG, Dalm VASH, Kootstra NA, Huckriede ALW, van Baarle D, Lafeber M, GeurtsvanKessel CH, de Vries RD, van der Kuy PM. Analyzing the immunogenicity of bivalent booster vaccinations in healthcare workers: The SWITCH ON trial protocol. Front Immunol. 2022 Nov 29;13:1067749. doi: 10.3389/fimmu.2022.1067749. eCollection 2022. PMID 36524126